CLINICAL TRIAL: NCT04885049
Title: A Randomized Controlled Trial Comparing the Efficacy of Anti Secretory and Oral Immunoglobulins Reducing the Episodes of Diarrhea in Children
Brief Title: Comparing the Efficacy of Anti-secretory Versus Oral Immunoglobulins for Reducing the Episodes of Diarrhea in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Nighat Haider, Assistant Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.F.1-1/2015/ERB/SZABMU/556
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — racecadotril; Suspensions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A (GA) will receive anti secretory 1.5mg/kg/dose three doses per oral in 24 hours for 3 days along with oral rehydration
  Interventions: Drug: Racecadotril
- Group B (Experimental): Group B (GB) will receive a single dose of bovine colostrum and egg solids as 7 g of dry powder reconstituted in 30 mL of water and taken orally once daily for 3 days along with oral rehydration
  Interventions: Drug: DiaResQ Children's Powder for Suspension

INTERVENTIONS:
Drug: Racecadotril — Anti secretary
  Arms: Group A
Drug: DiaResQ Children's Powder for Suspension — oral immunoglobulins
  Arms: Group B

SUMMARY:
Children 1-12 years presenting/admitted with acute diarrhea will be enrolled in the study after taking informed consent from the parents. Patients will be randomly allocated to two equal groups. Group A (GA) will receive anti secretory 1.5mg/kg/dose, three doses in 24 hours along with oral rehydration, while Group B (GB) will receive a single dose of bovine immunoglobulins. Response to treatment will be assessed by recording the frequency of loose stools after 72 hrs. Data will be collected through a structured proforma.

DETAILED DESCRIPTION:
It is a randomized clinical trial that will be conducted at Children Hospital PIMS, Islamabad over the period of 6 months. Sample size is calculated using World Health Organization (WHO) calculator, keeping confidence level 95%, level of significance 5%, power of the test 80%,anticipated population proportion 1: 84%, anticipated population proportion 2: 93%, which turn out to be 30.Consecutive non probability sampling technique will be used. Children 1-12 years both male and female visiting/admitted in Children Hospital PIMS with acute diarrhea of less than 15 days duration will be enrolled in the study after taking informed consent from the parents. Children requiring emergency resuscitation, having chronic diarrhea i-e more than 15 days duration, having other comorbid conditions like heart, kidney and liver failure, having metabolic disorder and who are allergic to egg or any of the contents will be excluded from the study.

Child's name, age, sex will be recorded by the on duty doctor. Patients will be randomly allocated to two equal groups. Group A (GA) will receive anti secretory 1.5mg/kg/dose three doses per oral in 24 hours along with oral rehydration, while Group B (GB) will receive a single dose of bovine colostrum and egg solids as 7 g of dry powder reconstituted in 30 mL of water and taken orally once daily for 3 days along with oral rehydration. Response to treatment will be assessed by recording the reduction in frequency of diarrheal episodes after administration of drug and duration in which the diarrheal episodes were reduced. Data will be collected through a structured proforma.

All data will be analyzed using latest SPSS version. Quantitative variables such as age, time will be presented as means and standard deviations. Qualitative variables such as age groups, sex, recurrence of seizures and efficacy will be measured as frequency and percentages. Effect modifiers like age, gender will be controlled by stratification. Post stratification chi-square test will be applied keeping p value ≤0.05 as significant.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-12 years both male and female visiting/admitted in Children Hospital PIMS with acute diarrhea of less than 15 days duration

Exclusion Criteria:

* Children requiring emergency resuscitation.
* Children having diarrhea of more than 15 days duration..
* Children with other comorbid conditions like heart, kidney and liver failure.
* Children with fructose intolerance, glucose malabsorption syndrome and saccharase isomaltase deficiency.
* Children allergic to egg or any of the contents.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
frequency of diarrheal episodes | 24 to 72 hours
  reduction in frequency of diarrheal episodes after administration of drug

CONTACTS AND LOCATIONS:
Overall Officials: Nighat Haider, FCPS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University

IPD SHARING:
Plan to Share IPD: Yes
If somebody wants the IPD they can email the principal investigator and it will be provided after the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of data.
Access Criteria: If somebody wants the IPD they can email the principal investigator and it will be provided